CLINICAL TRIAL: NCT00880477
Title: Immunogenicity and Safety of GSK Biological's DTPa-HBV-IPV/Hib Vaccine or DTPa-IPV/Hib Co-administered With HBV Vaccine as Primary and Booster Vaccination in Healthy Infants Born to Hepatitis B Surface Antigen Negative Mothers
Brief Title: Immunogenicity and Safety of Primary and Booster Vaccination With DTPa-HBV-IPV/Hib Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 217744/069
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: DTPa-HBV-IPV/Hib vaccine
- Group B (Experimental)
  Interventions: Biological: DTPa-IPV/Hib vaccine; Biological: EngerixTM-B

INTERVENTIONS:
Biological: DTPa-HBV-IPV/Hib vaccine — Vaccination according to a 3-dose schedule at 1 ½, 3 ½ and 6 months of age with booster at 15-18 months of age.
  Arms: Group A
Biological: DTPa-IPV/Hib vaccine — Vaccination according to a 3-dose schedule at at 1 ½, 3 ½ and 6 months of age with booster at 15-18 months of age.
  Arms: Group B
Biological: EngerixTM-B — The vaccine was administered according to a 2-dose schedule at 1½ and 6 months of age with booster at 15-18 months of age.
  Arms: Group B

SUMMARY:
This study will assess the immunogenicity, safety and reactogenicity of GSK Biological's DTPa-HBV-IPV/ Hib vaccine as compared to GSK's DTPa-IPV/Hib vaccine co-administered with HBV according to a three-dose immunisation course and as a booster dose in infants born to hepatitis B antigen seronegative mothers and previously primed with a birth dose of GSK's HBV vaccine.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for enrolment at birth

* Written informed consent obtained from the parents or guardians of the subject.
* A male or female infant born after a normal gestation period (between 36 and 42 weeks).
* Born to a mother seronegative for HBsAg.
* Free of obvious health problems as established by clinical examination before entering into the study.

Inclusion criteria for administration of the combined vaccine regimen

* Between, and including, 6 and 8 weeks of age at the time of the first dose of the three-dose course of vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into this phase of the study.

Inclusion criteria for administration of the booster dose

* Between, and including, 15 and 18 months of age at the time of the booster vaccination.
* Written informed consent obtained from the parents or guardians of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Completion of the three-dose primary vaccination course.

Exclusion Criteria:

Exclusion criteria for enrolment at birth

* A family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection.
* Major congenital defect(s).

Exclusion criteria for administration of the combined vaccine regimen

* Use of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration Immunosuppressants or other immune-modifying drugs since birth.
* Any chronic drug therapy to be continued during the study period.
* Planned administration/ administration of a vaccine except Bacille Calmette-Guérin vaccine during the period starting from 30 days before each dose of vaccines and ending 30 days after.
* Previous vaccination against diphtheria, tetanus, pertussis or Haemophilus influenzae type b disease.
* History of, or intercurrent, diphtheria, tetanus, pertussis, hepatitis B and/or Haemophilus influenzae type b disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Exclusion criteria for administration of the booster dose

* Use of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding the booster dose of study vaccines, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months of vaccination.
* Previous booster vaccination against diphtheria, tetanus, pertussis, hepatitis B, polio and/or Haemophilus influenzae type b.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* History of any neurologic disorders or seizures.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster dose of study vaccine or planned administration during the study period.
* Hypersensitivity reaction due to vaccine in primary course
* Encephalopathy within 7 days of previous vaccination with DTP vaccine

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2001-01; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Seroprotective anti-HBs antibody titres above protocol specified cut-off value | At the time of the second dose of combined vaccination, one month after the 3rd dose of combined vaccination and one month after the booster dose.

SECONDARY OUTCOMES:
Antibody titres against all investigational vaccine antigen components | One month after first combined vaccine dose, two months after Dose 1, one month after third combined vaccine dose prior to booster vaccination and one month post-booster vaccination.
Occurrence of solicited symptoms | During the 4-day follow-up period after each dose
Occurrence of unsolicited symptoms | During the 30-day follow-up period after each dose of study vaccine
Occurrence of Serious Adverse Events | From the birth dose of hepatitis B vaccine and ending with the last study visit or performance of the last study procedure or a minimum of 30 days following the third dose of the mixed vaccines and from the start of booster dose and ending a minimum of 3

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Shao PL, Lu CY, Hsieh YC, Bock HL, Huang LM; Taiwan Infanrix-069 Study Group. Immunogenicity and reactogenicity of DTPa-IPV/Hib vaccine co-administered with hepatitis B vaccine for primary and booster vaccination of Taiwanese infants. J Formos Med Assoc. 2011 Jun;110(6):415-22. doi: 10.1016/S0929-6646(11)60061-2. PMID 21741011
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 217744/069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 217744/069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 217744/069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 217744/069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 217744/069 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register